CLINICAL TRIAL: NCT03928535
Title: Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in Patients With Hypercapnic COPD，a Randomized Controlled Trial
Brief Title: Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation in Patients With Hypercapnic COPD
Acronym: COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 261358454
Record Dates: First submitted 2019-04-13; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2018-12

CONDITIONS: High-Flow Nasal Cannula; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Flow Nasal Cannula (Other): High-flow oxygen was applied immediately after extubation through specific nasal cannula.
  Interventions: Device: High-FlowNasal Cannula
- Noninvasive Ventilation (Other): Noninvasive Ventilation was applied immediately after extubation.
  Interventions: Device: Noninvasive Ventilation

INTERVENTIONS:
Device: High-FlowNasal Cannula — High-flowoxygenwas applied immediately after extubation through specific nasal cannula. Flow was initially set at 10 L/min and titrated upwards in 5-L/min steps until patients experienced discomfort.Temperature was initially set to 37°C, unless reported too hot by patients, and FIO2 was regularly adjusted to the target peripheral capillary oxygen saturation (SPO2) of greater than 92%. After 24 hours, high-flow was stopped and, if necessary, patients received conventional oxygen therapy.
  Arms: High-Flow Nasal Cannula
Device: Noninvasive Ventilation — Full face mask NIV was continuously delivered immediately after extubation for a scheduled period of 24 hours after extubation. Afterward, NIV was withdrawn and oxygen was administered by Venturi mask.Both PEEP and inspiratory pressure supportwere adjusted to target a respiratory rate of 25/min and adequate gas exchange (arterial oxygen saturation [SaO2] 92%, with pH of 7.35). The FIO2 was adjusted to maintain SPO2 at less than 92%. Sedatives to increase tolerance to NIV were not allowed.
  Arms: Noninvasive Ventilation

SUMMARY:
To test if high-flow conditioned oxygen therapy is noninferior to NIV for preventing postextubation respiratory failure and reintubation in patients with hypercapnic COPD, investigators plan to conduct the participants level, 1:1 randomized trial at the respiratory ICU. Participants were randomized to undergo either high-flow conditioned oxygen therapy or noninvasive mechanical ventilation after extubation. Primary outcomes were reintubation and postextubation respiratory failure within 72 hours. Secondary outcomes included length of RICU stay after extubation and mortality; partial pressure of arterial carbon dioxide.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AECOPD
* Extubation must be performed after 48 hours of invasive ventilation
* Must be treated sequentially with HFNC or NIV after extubation
* PaCO2≥50mmHg when extubation
* Positive End Expiratory Pressure (PEEP) ≤8cmH2O (1cmH2O=0.098 kPa) when extubation

Exclusion Criteria:

* Do-not-intubate
* Tracheostomies
* Accidental extubation
* Self-extubation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of reintubation | Within 72 hours after extubation
  The proportion of patients requiring reintubation within 72 hours after extubation

SECONDARY OUTCOMES:
RICU length of stay after extubation | From date of extubation until the date of discharging from the RICU up to 28 days
  Length of time from extubation to discharging from the RICU
Mortality | Within 28 days after extubation
  Mortality after extubation
Partial pressure of arterial carbon dioxide | Within 24 hours before extubation and within 72 hours after extubation
  Partial pressure of arterial carbon dioxide tested at the appointed time

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided